CLINICAL TRIAL: NCT04653844
Title: SARS-Cov2 (COVID-19) Infection and Reinfection Through the Analysis of a RT-PCR Results Database
Brief Title: RT-PCR Database Analysis for COVID-19 Infections and Re-infection
Acronym: ReCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Laboratoire CERBA-MPL (Unknown); CNRS (MIVEGEC) (Unknown); Nîmes University Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0640
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Covid-19; SARS-CoV Infection
Keywords: SARS-Cov2 infection; Positive SARS-Cov2 RT-PCR; SARS-Cov2 immune status; reinfection; kinetics; Rt-PCR; immunity
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Reinfection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SARS-Cov2 pandemic remains associated with many concerns. One of the them is the real frequency of likely re-infection and subsequently the level of protection conferred by the acquired immunity following primary-infection. We propose to analyze a large set of laboratory data produced since the early beginning of the SARS-Cov2 spread in the French population to identify recurrent infection events and, more generally, gain insight about infection kinetics.

ELIGIBILITY:
Inclusion criteria:

- People with at least one positive SARS-Cov2 RT-PCR result with a known sampling date

Exclusion criteria:

- Patient refusing to participate in research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: French population with a positive SARS-Cov2 diagnosis documented through a positive RT-PCR result
Sampling Method: Non-Probability Sample
Enrollment: 7000000 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 reinfection rate | 1 day
  SARS-CoV-2 reinfection rate

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Foulongne, PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC